CLINICAL TRIAL: NCT04210934
Title: Study of the Feature of Intestinal Microbiota and Its Role in Healthy Aging in Southern Chinese From a Longevity County, Yongfu
Brief Title: Study of Microbiota in Longevity County, Yongfu
Acronym: SoMiLY
Status: Completed | Type: Observational
Sponsor: Beijing Hospital (Other Government)
Collaborators: BGI-Shenzhen (Industry)
Responsible Party: Principal Investigator, Liang Sun, PhD, Director of Department of Medical Genetics, Beijing Hospital
Other Study IDs: 20170307
Record Dates: First submitted 2019-12-22; First posted 2019-12-26 (Actual); Last update posted 2019-12-27 (Actual); Status verified 2019-12

CONDITIONS: Aging; Healthy Aging
Keywords: Microbiota; multi-omics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — peripheral blood blood, 2 mL (serum) faeces, 200 mg
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is an observational study designed to adopt a cross-sectional study design. In the context of China's longevity town (East Asian population), Yongfu, Guangxi, the background of non-medical care and antibiotic use was explored, and the intestinal microecological balance increased with age and natural health. Longevity relationship. This study was completed using a household survey. Through routine clinical examinations and analysis of biochemical laboratory indicators, at the same time, a questionnaire for ADL(activities of daily living), cognitive function, and related elderly information was carried out on the elderly to comprehensively provide health information for each elderly. Based on the remaining stool samples and serum samples, the second-generation sequencing technology and other omics-based technologies were explored. No additional collection of human specimens and information is involved.

In addition, this study also hopes to explore the transmission rules of age-related bacteria in long-lived families, and the relationship with health phenotypes such as blood sugar, blood lipids, and cognitive function. Potential impact. In summary, this study will provide data support for exploring the relationship between healthy longevity and intestinal microecological balance based on the characteristic population of the longevity hometown.

ELIGIBILITY:
Inclusion Criteria:

* Obtained informed consent signed by volunteer or guardian
* Local lived for more than 50 years

Exclusion Criteria:

* Subjects being treated with antibiotic in 3 months
* People who cannot cooperate with completing the survey
* Severe gastrointestinal disorders

Ages: 22 Years to 111 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The current study was based on the Longevity and Health of Aging Population in Guangxi China (LHAPGC) study conducted in Yongfu County (qualified as the longevity town by Geriatric Society of China) in 2016.The enrolled subjects do not rely on medical care and do not take antibiotics recently. They are representative of a natural healthy-aging population model .
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2016-05-22 (Actual); Primary Completion 2016-05-31 (Actual); Study Completion 2016-05-31 (Actual)

PRIMARY OUTCOMES:
Aging-related fecal microbiota annotation | 0 week
  Taxonomy of bacteria(family,genus,species),Gene of bacteria

SECONDARY OUTCOMES:
interface of microbiota and other biomarkers in aging and related conditions | 0 week
  to study the correlation between microbiota and circulating biomarkers, including metabolite, and the shifts in various aging and related conditions

CONTACTS AND LOCATIONS:
Overall Officials: Liang Sun, Ph.D., Principal Investigator — Beijing Hospital; Ze Yang, M.D., Study Director — Beijing Hospital

IPD SHARING:
Plan to Share IPD: Undecided